CLINICAL TRIAL: NCT06723444
Title: Testing the Efficacy of a Memory Training Program to Improve New Learning and Memory in Portuguese Patients With Multiple Sclerosis: A Randomized Clinical Trial
Brief Title: Improving Learning and Memory in Portuguese Patients With Multiple Sclerosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centro Hospitalar De São João, E.P.E. (Other)
Collaborators: Instituto de Saude Publica da Universidade do Porto (Other); Center of Psychology at University of Porto (Unknown)
Responsible Party: Principal Investigator, Márcia Inês Teixeira França, Psychologist, Centro Hospitalar De São João, E.P.E.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CE-54-2024; 2024.05693.BDANA (Other Grant/Funding Number: Fundação para a Ciência e Tecnologia)
Record Dates: First submitted 2024-11-15; First posted 2024-12-09 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Memory; Cognitive Rehabilitation; Randomized Controlled Trial
MeSH Terms: conditions — Multiple Sclerosis | interventions — Educational Status; Cognitive Training

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The intervention group will receive paper and pencil learning and memory training exercises, administered twice a week for five weeks (10 training sessions).
  Interventions: Behavioral: Learning and Memory Training
- Placebo Control Group (Placebo Comparator): The placebo control group will receive paper and pencil placebo memory exercises administered twice a week for five weeks (10 placebo control sessions).
  Interventions: Behavioral: Placebo Comparator

INTERVENTIONS:
Behavioral: Learning and Memory Training — The intervention group will receive learning and memory retraining exercises, in order to learn how to apply two techniques: imagery and context.
  Paper and pencil memory retraining exercises will be administered twice a week for five weeks (10 training sessions).
  Arms: Intervention Group
Behavioral: Placebo Comparator — The placebo control group will receive paper and pencil placebo memory exercises, without learning techniques, administered twice a week for five weeks (10 placebo control sessions).
  Arms: Placebo Control Group

SUMMARY:
Deficits in memory and learning are common in Multiple Sclerosis, posing significant challenges in patients' daily lives. Cognitive rehabilitation has been shown to be effective in ameliorating these deficits, with programs such as the Modified Story Memory Technique (mSMT). In Portugal, no studies tested the efficacy of memory training programs. We aim to fill that gap by translating and developing mSMT, conducting a randomized double-blind, placebo-control, clinical trial, and, therefore, testing its efficacy through objective measures of cognitive function, and the maintenance of its benefits longitudinally. Patients with documented impairment in new learning abilities will be recruited at Centro Hospitalar Universitario São João, and randomly assigned to a memory retraining group or an active control group. Both groups will undergo baseline, immediate, and long-term follow-up assessments consisting of (1) a neuropsychological comprehensive assessment and (2) self-reported questionnaires regarding symptoms of anxiety, depression, fatigue, quality of life, and sleep. Optional enrollment in pre-post neuroimaging will also allow us to look at changes in the brain.

DETAILED DESCRIPTION:
Cognitive impairment in Multiple Sclerosis (MS) can manifest insidiously even before other neurological symptoms, with 40% to 65% of patients experiencing deficits. Long-term memory is consistently affected, with weak initial learning tending to lead to poor retrieval. Despite being invisible, cognitive problems in MS present significant challenges, as pharmacological treatments have shown limited efficacy in improving cognitive functions. Meanwhile, cognitive rehabilitation proves beneficial and meaningful among MS patients, with optimal outcomes observed at early stages.

The modified Story Memory Technique (mSMT) aims to ameliorate learning and memory deficits and has proven to be effective throughout three realms of assessment: objective cognitive abilities, daily life functioning, and neuroimaging. Its efficacy was already tested in different populations namely MS, progressive MS only, and traumatic brain injury. The mSMT involves ten individual sessions conducted twice weekly over five weeks, incorporating techniques such as imagery, context, and generalization. In the first four sessions, participants read stories for which they must create visual imagery to aid memory - imagery. In sessions 5 to 8, participants have word lists that they embed in a story and then visualize it - context. Sessions 9 and 10 apply mSMT to real-world situations (e.g., directions, to-do lists, and shopping) - generalization. Booster sessions may also be administered to maintain treatment effects over time. Previous studies have shown that memory improvements were sustained even six months after completion, highlighting its efficacy in MS. Neuroimaging studies proved the clinical utility of this intervention with significant changes in cerebral activation in regions associated with imagery and verbal learning, results considered extremely promising for the field of neurorehabilitation. Recognizing the need for cognitive rehabilitation programs adapted to Portuguese MS patients, the main objective of this project is to develop and test the efficacy of the Portuguese version of mSMT on MS patients in a hospital setting. This will be done through a Randomized Clinical Trial (RCT) throughout three realms of assessment: behavioral, neuropsychological, and neuroimaging.

Aim 1. Test the efficacy and the clinical utility of the Portuguese version of mSMT through objective measures of cognitive function and self-reported questionnaires regarding symptoms of anxiety, depression, fatigue, quality of life, and sleep. For this purpose, we will conduct a randomized double-blind, placebo-control, clinical trial in a hospital setting.

Aim 2. Assess the efficacy of this memory retraining protocol in a mildly impaired group and a moderate to severely impaired group.

Aim 3. Examine the maintenance of treatment effects longitudinally, through the inclusion of 6-month and 18-month follow-up assessments.

Aim 4. Examine the mSMT efficacy considering variables such as the previous neuropsychological profile and neuroimaging data.

ELIGIBILITY:
Inclusion Criteria:

* established diagnosis of MS, according to McDonald criteria;
* adult native Portuguese speakers;
* at least four years of education;
* free of exacerbations and use of steroids for at least one month, and no neurologic history other than MS;
* no history of major depressive disorder, schizophrenia, bipolar disorder, and no history of substance use/dependence;
* no significant visual impairment that impacts the ability to see testing materials and language comprehension as measured by the Token Test;
* impaired verbal new learning as documented by a performance of -1.0 or worse standard deviations below the mean, using age, sex and education-adjusted Portuguese norms on the Selective Reminding Test from the Brief Repeatable Battery of Neuropsychological Tests.

Exclusion Criteria:

* an exacerbation within one month;
* neurological history of head injury, stroke, seizures, or any other significant neurological history;
* patients on steroids, benzodiazepines, and/or neuroleptics;
* patients with an active diagnosis of Major Depressive Disorder, Schizophrenia, Bipolar Disorder;
* poor visual acuity, diplopia, or nystagmus;
* inability to understand directions and following one, two, and three step commands;
* and intact new learning and memory.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-12-05 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Verbal memory | Four points in time: pre-treatment, immediately following treatment, 6 months and 18 months after treatment is completed.
  Selective Reminding Test from Brief Repeatable Battery of Neuropsychological Tests (BRBN-T), with higher scores mean better outcome performance.
Verbal memory | Four points in time: pre-treatment, immediately following treatment, 6 months and 18 months after treatment is completed.
  California Verbal Learning Test II from Brief International Cognitive Assessment for Multiple Sclerosis (BICAMS), with higher scores mean better outcome performance.

SECONDARY OUTCOMES:
Self-reported Questionnaires | Four points in time: pre-treatment, immediately following treatment, 6 months and 18 months after treatment is completed.
  Hospital Anxiety and Depression Scale (HADS), a self-assessed questionnaire consisting of 14 items (0-3 Likert scale) assessing symptoms of depression (HADS-D subscale) and anxiety (HADS-A subscale).
Self-reported Questionnaires | Four points in time: pre-treatment, immediately following treatment, 6 months and 18 months after treatment is completed.
  Modified Fatigue Impact Scale (MFIS), with a score range of 0-84 for each item, with the highest score indicating greater fatigue severity.

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Hospitalar Universitário de São João, Porto, Portugal